CLINICAL TRIAL: NCT02315729
Title: Analysis of Prognostic Cell Signaling Factors in Adolescent Idiopathic Scoliosis
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0884; UL1TR001082 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to identify potential markers for curve progression in adolescent idiopathic scoliosis (AIS). Despite its prevalence and impact on child health, the etiology of AIS and molecular mechanisms underlying its development and progression remain poorly understood. Clinical criteria and features cannot adequately predict which children, diagnosed with mild disease, will undergo subsequent curve progression requiring intervention.

The investigators hypothesize that alterations in specific genetic markers will be correlated with the progression of AIS curves over time. Thus, these markers could be used in the future to develop a reliable, inexpensive and relatively non-invasive cell based diagnostic test to (1) predict spinal curve progression in AIS, (2) select patients likely to benefit from early surgical intervention, and (3) potentially screen for asymptomatic children at risk of developing idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 10-13 years
* Diagnosed with mild-moderate spine deformity (Cobb angle 15-30 degrees)

Exclusion Criteria:

* Patients with scoliosis other than idiopathic
* Trauma
* Inflammatory disease
* Malignancies
* Diabetes
* History of previous spine surgery

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Female patients with adolescent idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2016-11; Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Progression | 3 years
  Cobb angle, disc wedging, vertebral body wedging, coronal balance, sagittal balance

CONTACTS AND LOCATIONS:
Overall Officials: Evalina L Burger, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children'S Hospital of Colorado, Denver, Colorado, United States